CLINICAL TRIAL: NCT01803269
Title: A Randomized Phase II Study of IV Topotecan Versus CRLX101 in the Second Line Treatment of Recurrent Small Cell Lung Cancer
Brief Title: Topotecan Hydrochloride or Cyclodextrin-Based Polymer-Camptothecin CRLX101 in Treating Patients With Recurrent Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lack of activity and slow accrual
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-1726; NCI-2013-00402 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-27; First posted 2013-03-04 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-04

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan; trioctyl phosphine oxide; IT-101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (topotecan hydrochloride) (Active Comparator): Patients receive topotecan hydrochloride IV over 30 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: topotecan hydrochloride
- Arm B (CRLX101) (Experimental): Patients receive cyclodextrin-based polymer-camptothecin CRLX10 cyclodextr1 IV over 60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclodextrin-based polymer-camptothecin CRLX101

INTERVENTIONS:
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
  Arms: Arm A (topotecan hydrochloride)
Drug: cyclodextrin-based polymer-camptothecin CRLX101 — Given IV
  Other Names: CRLX101; cyclodextrin-based polymer-camptothecin IT-101; IT-101
  Arms: Arm B (CRLX101)

SUMMARY:
This randomized phase II trial studies how well giving topotecan hydrochloride or cyclodextrin-based polymer-camptothecin CRLX101 works in treating patients with recurrent small cell lung cancer. Drugs used in chemotherapy, such as topotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Cyclodextrin-based polymer-camptothecin CRLX101 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet know whether topotecan hydrochloride is more effective than cyclodextrin-based polymer-camptothecin CRLX101 in treating patients with lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of second-line treatment with CRLX101 (cyclodextrin-based polymer-camptothecin CRLX101) compared to intravenous (IV) topotecan hydrochloride (topotecan) on progression free survival (PFS) of patients with extensive-stage small cell lung cancer (ES-SCLC) sensitive to first-line platinum-based chemotherapy.

II. To evaluate the effect of second-line treatment with CRLX101 on the three-month PFS rate of patients with ES-SCLC resistant to first-line platinum-based chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate the response rate of second-line treatment with CRLX101 in patients with ES-SCLC who are sensitive or resistant to first-line platinum-based chemotherapy.

II. To evaluate the effect of second-line treatment with CRLX101 compared to IV topotecan on overall survival (OS) of patients with ES-SCLC sensitive to first-line platinum-based chemotherapy.

III. To assess the overall survival of second-line treatment with CRLX101 in patients with ES-SCLC resistant to first-line platinum-based chemotherapy.

IV. To assess the toxicity of second-line CRLX101 in patients sensitive or resistant to first-line platinum-based chemotherapy.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A (Sensitive Relapse): Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive topotecan hydrochloride intravenously (IV) over 30 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive cyclodextrin-based polymer-camptothecin CRLX101 IV over 60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

COHORT B (Resistant Relapse): Patients receive cyclodextrin-based polymer-camptothecin CRLX101 as in Arm B Cohort A. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed small cell lung cancer

  * All patients must have extensive stage disease; extensive stage patients are defined as those patients with bilateral or contralateral supraclavicular adenopathy or contralateral hilar adenopathy or malignant pleural effusion or extrathoracic metastatic disease
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients must have been treated with 1 prior platinum-based (cisplatin or carboplatin) regimen; prior thoracic radiation for limited stage disease is allowed; patients must be at least 4 weeks since prior chemotherapy or radiation
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Baseline imaging studies performed =< 28 days of study registration
* The effects of CRLX101 on the developing human fetus are unknown; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of CRLX101 administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who have previously been treated with irinotecan or topotecan
* Patients who are receiving any other investigational agents
* Patients with uncontrolled brain metastases; patients with treated brain metastases must have stable neurologic status off of steroids and anticonvulsants for at least 2 weeks and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CRLX101 or topotecan
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Previous or concurrent malignancy; exceptions: treated basal cell or squamous cell skin cancer, in situ cervical cancer, or lobular carcinoma in situ in one breast; or other cancer which the patient has been disease-free >= 5 years
* Pregnant women and women who are capable of reproduction but who will not agree to use adequate contraception prior to study entry and for the duration of study participation; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CRLX101 or topotecan, breastfeeding should be discontinued if the mother is treated with either agent
* Human immunodeficiency virus (HIV)-positive patients
* Patients with history of inflammatory bowel disease requiring therapy or patients with chronic diarrhea syndromes or paralytic ileus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-01-16 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Salgia, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (5):
- United States (5):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - North Shore University Health System, Evanston, Illinois
  - Ingalls Memorial Hospital, Ingalls Park, Illinois
  - Illinois Cancer Care, Peoria, Illinois

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort C: Non-randomized group that had no response to 1st line therapy or relapse within 60 days after completion of first-line chemotherapy
Period: Overall Study
Arm/Group | Arm A (Topotecan Hydrochloride) | Arm B (CRLX101) | Cohort C
Started | 7 | 8 | 14
Completed | 4 | 8 | 14
Not Completed | 3 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Topotecan Hydrochloride) | Arm B (CRLX101) | Cohort C | Total
Number analyzed (Participants) | 7 | 8 | 14 | 29
Age, Continuous [Mean (Full Range); unit: years] | 68.9 [56 to 83] | 68.1 [52 to 80] | 67.3 [42 to 87] | 67.9 [42 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 7 | 13
  Male | 4 | 5 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 3 | 5
  White | 7 | 6 | 11 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Time from enrollment to disease progression or death from any cause
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Topotecan Hydrochloride) | Arm B (CRLX101) | Cohort C
Number analyzed (Participants) | 7 | 8 | 14
months | 1.3 [0.5 to 1.8] | 2.1 [0.7 to 2.9] | 1.3 [0.9 to 2.2]

2. Secondary Outcome: Response Rates According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (Cohort A)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Population: Patients initiating treatment (i.e., exclude 3 withdrawals prior to starting treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Topotecan Hydrochloride) | Arm B (CRLX101) | Cohort C
Number analyzed (Participants) | 4 | 7 | 11
Participants | 1 | 0 | 0

3. Secondary Outcome: Continuous Change in Tumor Size.
Description: Change in sum of longest diameters of all target lesions from baseline to end of cycle 2.
Time Frame: Up to 56 days
Population: Patients completing two cycles of therapy.
Measure: Mean (Standard Error); unit: mm
Arm/Group | Arm A (Topotecan Hydrochloride) | Arm B (CRLX101) | Cohort C
Number analyzed (Participants) | 2 | 7 | 9
mm | -50.0 (42.0) | 16.8 (6.1) | 5.1 (6.1)

4. Secondary Outcome: Overall Survival
Description: Time from enrollment until death from any cause
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Topotecan Hydrochloride) | Arm B (CRLX101) | Cohort C
Number analyzed (Participants) | 7 | 8 | 14
months | 4.0 [0.5 to 20] | 5.3 [2.0 to 12.5] | 2.5 [1.2 to 7.3]

5. Secondary Outcome: Frequency of Reported Side Effects
Description: Any adverse event regardless of grade or attribution
Time Frame: Up to 3 years after completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Topotecan Hydrochloride) | Arm B (CRLX101) | Cohort C
Number analyzed (Participants) | 7 | 8 | 14
Participants | 4 | 7 | 12

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Arm A (Topotecan Hydrochloride) | Arm B (CRLX101) | Cohort C
All-Cause Mortality (participants affected / at risk) | 3/7 | 8/8 | 14/14
Serious Adverse Events (participants affected / at risk) | 3/7 | 3/8 | 5/14
Other Adverse Events (participants affected / at risk) | 2/7 | 6/8 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Topotecan Hydrochloride) (N=7) | Arm B (CRLX101) (N=8) | Cohort C (N=14)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Death NOS (General disorders) | 1 | 0 | 2
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Hallucinations (Psychiatric disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Acute mental status change (Psychiatric disorders) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Topotecan Hydrochloride) (N=7) | Arm B (CRLX101) (N=8) | Cohort C (N=14)
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 2
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 4
Confusion (Psychiatric disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 5
Dysgeusia (Nervous system disorders) | 1 | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 7
Edema limbs (General disorders) | 1 | 2 | 3
Facial pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 8
Fever (General disorders) | 1 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 4
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Hypotension (Vascular disorders) | 1 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 2
Platelet count decreased (Investigations) | 2 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 1
Tremor (Nervous system disorders) | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
White blood cell decreased (Investigations) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Bloating (Gastrointestinal disorders) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 2
CD4 lymphocytes decreased (Investigations) | 0 | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 2
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Flu like symptoms (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 6
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Pain (General disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 0 | 2
Hallucinations (Psychiatric disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 3
Hot flashes (Vascular disorders) | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No